CLINICAL TRIAL: NCT00051805
Title: Promoting Adherence to Antiretroviral Regimens
Brief Title: Promoting Adherence to Anti-HIV Drug Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel
Other Study IDs: 1R01AI045403-01A2 (NIH); 3R01AI045403-02S1 (NIH); 5R01AI045403-03 (NIH); NCT00078780 (obsolete NCT alias)
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: Patient Compliance; Adherence; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Patient Compliance

INTERVENTIONS:
Behavioral: Promotion of adherence to ARV medications

SUMMARY:
One of the main causes of treatment failure in HIV infected individuals is lack of adherence to complicated drug regimens. The purpose of this study is to evaluate the effectiveness of a behavioral intervention program designed to improve adherence to anti-HIV drug regimens. Participants in this study will be recruited from the University of Alabama at Birmingham (UAB) Outpatient HIV Clinic.

DETAILED DESCRIPTION:
Poor adherence to complicated antiretroviral (ARV) drug regimens is one of the most pressing behavioral problems in the clinical management of HIV infected persons. Recent medical advances have made it possible to maintain tighter control of viral replication, allowing people with HIV to live longer, healthier lives. However, the complexity of ARV drug regimens and drug side effects make medication adherence problematic. Deviations from the prescribed regimen may allow the virus to resume rapid replication and develop drug resistant mutations that could render the prescribed drugs useless. This study will evaluate the efficacy of a 6-month, theory-based behavioral intervention to enhance adherence to antiretroviral treatment regimens. HIV-related attitudes, depressive symptoms, coping strategies, and social support will also be assessed to examine theoretical assumptions regarding the causal relationship between psychosocial constructs and medication adherence.

Participants in this study will be recruited from UAB Outpatient HIV Clinic patients who are taking ARV medication. Participants will be randomized to a Standard Adherence Promotion Group or an Enhanced Adherence Promotion Group. The Enhanced Adherence Promotion will systematically address specific psychosocial issues associated with medication adherence. Participants will be followed for 6 months, and adherence will be evaluated at monthly study visits. Pill counts, viral loads, self-reported adherence to ARV medication, CD4 count, and genotypic viral resistance will be assessed.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* Receiving services at UAB Outpatient HIV Clinic
* Taking antiretroviral medication
* Able to attend monthly assessment meetings at clinic for 6 months
* Passing score on Mini Mental State Examination

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119
Dates: Start 2002-08; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Pill counts for ARV medications

SECONDARY OUTCOMES:
Viral load
disease progression measures (CD4 count, viral resistance)
self-reported adherence
self-reported psychosocial measures

CONTACTS AND LOCATIONS:
Overall Officials: Polly Kratt, PhD, MSPH, Principal Investigator — University of Alabama at Birmingham Outpatient HIV Clinic
Locations (1):
- University of Alabama at Birmingham Outpatient HIV Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Background] Stewart KE,Greene PG,Ross D,Kratt P, Balentine C, Lee P, Wang Y. Sex, drugs, and viral load: Associations in an HIV+ cohort. In: Society of Behavioral Medicine, 27th Annual Meeting & Scientific Sessions; 2006 Mar 23; San Francisco [CA]: Behavioral Medicine Across the Lifespan. Session Abstracts & Program Information Vol. 31, No. suppl. 1, Pages i-I.